CLINICAL TRIAL: NCT06180499
Title: Allogeneic Immunotherapy of Hematological Malignancies Using Regulatory T-cell Selective Depletion
Acronym: ILDTreg2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P120103
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hematological Malignancies; Regulatory T Cell Depletion; Relapse
Keywords: DLI; Regulatory T cells depletion; Hematological malignancies; Relapse
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T-reg depleted DLI (Experimental)
  Interventions: Drug: T-reg depleted DLI

INTERVENTIONS:
Drug: T-reg depleted DLI — Treg depleted Donor Lymphocytes Infusion

SUMMARY:
Since the discovery that Treg suppress anti-tumor immune responses, inhibiting their function has become a major challenge for the development of efficient immunotherapy for cancer. In humans, we previously reported the positive results of a first clinical trial using Treg depletion for anti-tumor response amplification in the field of allogeneic hematopoietic stem cell transplantation (HSCT). The present project aims at developing this anti-tumor immunotherapeutic strategy in the same setting, i.e. donor lymphocyte infusion (DLI) for relapsing hematological malignancies after HSCT, using a new selection marker: CD127. The choice of this new strategy is supported by our results of a retrospective clinical study and pre-clinical data. Using human cells, this studies demonstrated, in vitro and in vivo in animal murine models, that Treg depletion through CD127 positive selection is much more efficient to improve allogeneic immune responses of donor T-cells as compared to the previous strategy using the CD25 marker.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (older than 18 years old without upper limit of age) diagnosed with leukemia, myelodysplasia, myeloproliferative disorder or lymphoproliferative disorder (CLL, myeloma, lymphoma)
* Previous allogeneic HSCT from a matched sibling, haplo-identical or unrelated donor (any type of conditioning regimen)
* Haematological relapse (molecular, cytogenetic or cytological) after HSCT
* Patient refractory (no or partial response) to one or several previous standard unmanipulated DLI
* Availability of cryopreserved lymphapheresis
* No loss of chance by using of DLI rather than more incisive anti-tumor agents according to investigator appreciation
* Written informed consent before any intervention necessary for the trial
* Affiliation to a social security regime
* Negative pregnancy test for women of childbearing age participating in the study
* Effective contraceptive methods for men / women in line with the current CTFG recommendations version 1.1

Exclusion Criteria:

* Acute grade ≥ II or moderate/severe chronic GVHD at the time of inclusion
* Patient receiving immunosuppressive treatment for GVHD or any other reason
* Creatinine clearance< 50 ml/min
* Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 5.0 x upper limit of normal (ULN)
* Serum total bilirubin > 50µM (expect for unconjugated hyperbilirubinemia due to Gilbert's disease)
* Performance status ECOG>1
* Severe infection according to CTCAE grading (grade>2)
* Pregnant or lactating women
* Patient under tutorship, curatorship or legal protection
* Ongoing participation in another interventional research protocol within the same field of immune modulation (through cell therapy or not)
* State medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of GVHD in its acute grade ≥ II and/or severe chronic form (according Glucksberg-Thomas and NIH scales, respectively), and uncontrolled after a 14-day immunosuppressive course including steroids. | occurring within the 2 months following d-DLI infusion
  Composite criteria. In this evaluation, death from non-GVHD cause will be taken as a competitive event

SECONDARY OUTCOMES:
Incidence of acute and/or chronic GVHD, with corresponding grades according to NIH and Glucksberg-Thomas scales | at 2 and 12 month
Date of putative relapse/progression for estimation of cumulative incidence (taking into account the competitive risk of death not related to relapse) | at 2 and 12 month
Date of putative relapse/progression for estimation disease-free survival | at 2 and 12 month
Number, causes and date of deaths | at 2 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: elodie lemadre, M.Sc, Study Chair — APHP

IPD SHARING:
Plan to Share IPD: No